CLINICAL TRIAL: NCT01090622
Title: Phase 2a, Double-blind, Placebo-controlled, 2-period, Crossover Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Multiple Oral Doses of XPF-001 in Patients With Inherited Erythromelalgia.
Brief Title: Study of XPF-001 in the Treatment of Pain From Primary/Inherited Erythromelalgia (IEM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-001-202; 2009-015619-42 (EudraCT Number)
Record Dates: First submitted 2010-03-17; First posted 2010-03-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Primary Erythromelalgia; Inherited Erythromelalgia
MeSH Terms: conditions — Erythromelalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- XPF-001 (Experimental)
  Interventions: Drug: XPF-001

INTERVENTIONS:
Drug: XPF-001 — Oral capsule
  Arms: XPF-001
Drug: Placebo — Oral capsule
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine whether XPF-001 is safe and effective in the treatment of pain caused by Inherited Erythromelalgia (IEM).

ELIGIBILITY:
Inclusion Criteria:

The study requires you to:

* Be18-75 years old
* Have inherited erythromelalgia
* Be experiencing pain caused by erythromelalgia (Moderate pain score 4/10)
* Be generally healthy (apart from your pain)
* Stop taking your usual pain medications for 9 days
* Not be pregnant or breast-feeding

Your role in the study includes:

* An out-patient screening visit
* 9-days/8 nights-in-patient treatment visit at Nijmegen Medical Center (where you will be closely monitored)
* A follow up phone call (after your return home)
* Taking the investigational medication daily
* Recording your pain levels daily during stay at the Medical Center.

Exclusion Criteria:

* Coexistent source of pain from other conditions
* Receiving professional psychological support for dealing with IEM
* Treatment for significant depression within 6 months of screening
* Active HIV, Hepatitis B or C
* Use of prescription or OTC medication between check-in and discharge
* Women who are pregnant, or lactating
* Not currently using adequate contraception
* Alcoholism or alcohol or substance abuse
* Presence or history of major psychiatric disturbance
* Unwilling or unable to comply with all dietary and activity restrictions
* Any other condition or finding that may pose undue risk for participation
* Use of any other investigational drug in the 60 days prior to dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference (PID) in each treatment period based on an 11-point Pain Intensity-NRS (where 0 = No pain and 10 = worst pain you can imagine) | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Clinical Research Centre at Radboud University Nijmegen Medical Center, Nijmegen, Netherlands